CLINICAL TRIAL: NCT00045019
Title: An International Field-Testing Study Of The Reliability And Validity Of A Patient Satisfaction Module (QLQ-SAT32) Assessing Cancer Patients' Perception Of The Quality Of Care Received Within The Hospital
Brief Title: Study to Assess Cancer Patients' Satisfaction With Hospital Quality of Care
Status: Completed | Type: Observational
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Other Study IDs: EORTC-15012; EORTC-15012 (Other: EORTC)
Record Dates: First submitted 2002-09-06; First posted 2003-01-27 (Estimated); Last update posted 2012-08-27 (Estimated); Status verified 2012-08

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- discharged cancer patients: patients discharged from a surgery or medical ward of oncology institutes in Belgium, France, Germany, Italy, Poland, Spain, Sweden, Taiwan and United Kingdom (as part of a larger psychometric validation study) were asked to rate there level of satisfaction, using the EORTC QLQ-SAT32.
  Interventions: Other: quality-of-life assessment

INTERVENTIONS:
Other: quality-of-life assessment — QLQ-C30 SAT32
  Other Names: QoL

SUMMARY:
RATIONALE: Questionnaires may help determine cancer patients' satisfaction with the quality of care they received in the hospital.

PURPOSE: Clinical trial to determine the effectiveness of questionnaires in assessing cancer patients' satisfaction with the quality of care they received in the hospital.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the scale structure, reliability, and validity of the QLQ-SAT32 patient satisfaction module in assessing the perception of the quality of care received in hospitals by patients with cancer.
* Determine the success of the QLQ-SAT32 patient satisfaction module when used with the QLQ-C30 core quality of life questionnaire, in terms of expanding on quality of life evaluation or providing information on treatment acceptability or preference of these patients.

OUTLINE: This is a descriptive, multicenter study. Patients are stratified according to age (18 to 49 vs 50 and over) and the cancer therapy received in hospital (surgery vs chemotherapy).

Patients in all strata receive the QLQ-SAT32 and QLQ-C30 questionnaires, a debriefing questionnaire, and the Oberst patient satisfaction visual analog scale prior to hospital discharge. Patients complete the materials at home within 7 days of discharge. A group of 100 patients have a repeat QLQ-SAT32 module mailed to them to be completed within 7 days of receipt of first questionnaire.

PROJECTED ACCRUAL: A total of 640-768 patients (160-192 per stratum) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed cancer
* Hospitalization of at least 3 days
* No clinical evidence of brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* No psychological, familial, sociological, or geographical condition that would preclude study
* Able to understand the language of the questionnaire
* Mentally fit to complete a questionnaire

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Prior chemotherapy allowed

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Prior surgery for cancer allowed

Other

* No concurrent participation in other quality of life studies that would preclude this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cancer patients discharged from a surgery or medical ward of oncology institute.
Sampling Method: Non-Probability Sample
Enrollment: 795 (Actual)
Dates: Start 2002-05; Primary Completion 2004-06 (Actual); Study Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Bredart, Study Chair — Institut Curie
Locations (11):
- Institut Jules Bordet, Brussels, Belgium
- France (6):
  - Institut Bergonie, Bordeaux
  - Centre Regional Francois Baclesse, Caen
  - Institut Curie - Section Medicale, Paris
  - Centre Paul Strauss, Strasbourg
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif
- Hospital De Navarra, Pamplona, Spain
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg
  - Uppsala University Hospital, Uppsala
- Bristol Royal Infirmary, Bristol, United Kingdom